CLINICAL TRIAL: NCT00187174
Title: Phase I Trial of RAD001C (Everolimus) in Pediatric Patients With Recurrent Refractory Solid Tumors or Brain Tumors
Brief Title: Everolimus for Treating Pediatric Patients With Recurrent or Refractory Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD001
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2009-12

CONDITIONS: Tumors; Brain Tumors; Rhabdomyosarcoma; Sarcoma, Soft Tissue
Keywords: Brain tumors; Soft Tissue Sarcomas; Refractory solid tumors; Recurrent or Refractory Rhabdomyosarcomatous Soft Tissue and Non-Rhabdomyosarcoma Soft Tissue Sarcomas
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Rhabdomyosarcoma; Sarcoma; Recurrence | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1 (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — The drug is given orally in 28 day courses.

SUMMARY:
Patients with recurrent or refractory solid tumors or brain tumors that are unresponsive to conventional therapy, or with no known effective therapy, will be treated. Experiments in the laboratory have shown the experimental drug RAD001C (RAD001, Everolimus) can prevent cells from multiplying. RAD001 is now being tested in diseases such as cancer, in which excessive cell multiplication needs to be stopped. The drug has been tested in adult cancer patients and has been well tolerated by subjects in these studies. It is experimental and, therefore, available in clinical trials.

DETAILED DESCRIPTION:
Although a Phase II portion of this study was planned, it was never initiated.

ELIGIBILITY:
Inclusion Criteria:

* Adequate performance status
* Adequate bone marrow, kidney, heart, and liver function

Exclusion Criteria:

* Must not be receiving concomitant anti-cancer treatment
* Must not be pregnant

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To find the highest dose of RAD001 that can be given to children with refractory or relapsing solid tumors, leukemias, or brain tumors without causing severe side effects | Within 30 days per subject

SECONDARY OUTCOMES:
To find out if there are changes in the body's blood cells and tumor cells after treatment with RAD001 | Within 30 days per subject

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Furman, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org